CLINICAL TRIAL: NCT03539419
Title: Prospective Observational Study to Evaluate the Benefits for the Patient Associated With the Treatment of Plaque Psoriasis With Apremilast After Other Systemic Treatment in Conditions of Clinical Practice in Spain (APPROPRIATE Study)
Brief Title: Study to Evaluate the Benefits for the Patient Associated With the Treatment of Plaque Psoriasis With Apremilast After Other Systemic Treatment in Conditions of Clinical Practice in Spain
Acronym: APPROPIATE
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSOR-017; U1111-1212-0643 (Registry Identifier: WHO)
Record Dates: First submitted 2018-04-20; First posted 2018-05-29 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Psoriasis
Keywords: Psoriasis; Plaque Psoriasis; Apremilast; CC-10004
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with plaque psoriasis on apremilast: Adult patients with moderate to severe plaque who have started apremilast treatment for first time 3 months (+/- 4 weeks) before their inclusion in the study, according to the specifications of the drug's prescribing information and under usual clinical practice.

SUMMARY:
Observational, prospective and multicenter study in approximately 30 sites nationwide. The investigators participating in this study will be dermatologists specializing in this pathology.

The present study will include adult patients with moderate to severe plaque who have started apremilast treatment for first time 3 months (+/- 4 weeks) before their inclusion in the study, according to the specifications of the drug's prescribing information and under usual clinical practice. Recruitment will be consecutive and the reason for not including a potential candidate patient will be registered. The decision to prescribe apremilast treatment should be clearly dissociated from the inclusion of the patient in the study. Therefore, the choice of the therapeutic strategy will be made independently by the physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female (≥ 18 years).
* Patients diagnosed with moderate to severe plaque psoriasis and for which treatment with apremilast is indicated according to the doctor's criteria (established before the patient enters the study) and according to the specifications of the medication's data sheet
* Patients with available data regarding the PASI and DLQI assessments at the moment of initiating treatment with apremilast.
* Patients for whom, according to the physician's criteria (established prior to patient's entry into the study) and according to the specifications of the drug's prescribing information, apremilast treatment is indicated.
* All patients who, according to the routine clinical practice, initiated apremilast treatment for the first time 3 months (+/- 4 weeks) before their inclusion in the study (patients may or may not have completed 3 months of apremilast treatment).
* Patients who have previously received at least one systemic treatment for moderate to severe plaque psoriasis.
* Patients who have not previously been treated with a biological agent for moderate to severe plaque psoriasis.
* Patients who agree to participate in the study by signing the informed consent.
* Patients who are able to understand and complete the questionnaires specified in the study protocol.

Exclusion Criteria:

• Patients participating in another study at the time of entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients with moderate to severe plaque who have started apremilast treatment for first time 3 months (+/- 4 weeks) before their inclusion in the study, according to the specifications of the drug's prescribing information and under usual clinical practice. Recruitment will be consecutive and the reason for not including a potential candidate patient will be registered. The decision to prescribe apremilast treatment should be clearly dissociated from the inclusion of the patient in the study. Therefore, the choice of the therapeutic strategy will be made independently by the physician.
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving PBI ≥ 1 | Approximately 7 months
  Patient Benefit Index (PBI) is a measure of the benefit associated with a patient-reported treatment consisting of the administration of two questionnaires: the Patient needs questionnaire (PNQ), administered at baseline, and the patient benefit questionnaire (PBQ), administered during treatment

SECONDARY OUTCOMES:
Describe the persistence of apremilast treatment | Approximately 7 months
  Is defined as the duration of time from initiation to discontinuation of therapy.
Describe changes in the perception of pruritus intensity during apremilast treatment in patients with moderate to severe plaque psoriasis | Approximately 13 months
  Pruritus intensity measures: Usually used scales are based on patient perception: Visual analogue scale (VAS). Horizontal line of 100 mm, with descriptive signs at the ends indicating "no itching" and "the worst imaginable itch". The score is obtained by measuring the distance in millimeters from the beginning of the line to a vertical mark placed by the patient to indicate the intensity of the pain
Describe the changes in the quality of life associated with treatment with apremilast | Approximately 13 months
  The information on the variables studied will be obtained from the clinical record and the tests and evaluations carried out routinely during the patient follow-up who initiate a first treatment with apremilast, as well as the questionnaires for the evaluation of the dermatological quality of life (DLQI self-administered questionnaire), the evaluation of treatment satisfaction reported by the patient (PBI) and the intensity of pruritus (self-reported measures, VAS).
Describe the percentage of patients with moderate to severe plaque psoriasis who achieve a relevant minimum clinical benefit, defined as PBI ≥ 1 | Approximately 13 months
  Patient Benefit Index (PBI) is a measure of the benefit associated with a patient-reported treatment consisting of the administration of two questionnaires: the Patient needs questionnaire (PNQ), administered at baseline, and the patient benefit questionnaire (PBQ), administered during treatment.
Describe changes in concomitant medication associated with management of moderate to severe plaque psoriasis during apremilast treatment | Approximately 13 months
  Describe changes of concomitant medication specific for psoriasis associated to apremilast treatment indicating the date of beginning and end of the concomitant treatments that the patient receives during the treatment with apremilast.
Describe changes in cutaneous involvement of patients with psoriasis in severe intensity plaques that change to moderate intensity | Approximately 13 months
  A patient with moderate-intensity psoriasis will be considered if he/she has PASI 7-15 and DLQI scores ≤ 15, or PASI scores <7 and DLQI ≥ 5 at the time of starting apremilast treatment. (Patients with PASI 7-15 and DLQI> 15 scores and presenting cutaneous lesions in locations that are difficult to access for treatment or that have a significant psychosocial impact may be classified as moderate or severe psoriasis cases according to the investigators' criteria.) In this subgroup of patients will estimate the proportion of patients with moderate-intensity psoriasis who change to mild intensity.
Adverse Events (AEs) | Approximately 13 months
  Number of subjects with adverse event. Safety and tolerability to treatment will be assessed by the collection of adverse events (AE) occurring during follow-up.
Clinical and demographic characteristics of plaque psoriasis patients: Body surface affected (BSA). | Approximately 7 months
  Psoriasis is characterized as mild, moderate, or severe according to the amount of body surface area (BSA) affected and the severity of redness, thickness, and scaling of the skin. According to the centers usual clinical practice, the clinical assessment of psoriatic disease is based on the BSA. Percentage of body surface affected by psoriasis (scale 0-100).
Clinical and demographic characteristics of plaque psoriasis patients: Physician Global Assessment (PGA). | Approximately 7 months
  The Psoriasis Global Assessment (PGA) of improvement (or Physician's global assessment of improvement) measure the global assessment of the patient's overall severity of the disease on a 6-point scale, scored from "severe" to "clear".
Clinical and demographic characteristics of plaque psoriasis patients: PGA x BSA | Approximately 7 months
  Commonly used instruments for measuring psoriasis, such as Psoriasis Area and Severity Index (PASI), have limitations, including high complexity. PGAxBSA is a simple and sensitive instrument for measuring psoriasis severity. PGA×BSA is practical alternative to PASI for measuring severity and treatment response

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (53):
- Spain (53):
  - Hospital Juan Ramón Jiménez, Huelva, Andalusia
  - Complejo Hospitalario de Jaén, Jaén, Andalusia
  - Hospital Carlos Haya, Málaga, Andalusia
  - Research Site, Zaragoza, Aragon
  - Hospital Royo Vilanova, Zaragoza, Aragon
  - Hospital Dr Negrin, Las Palmas de Gran Canaria, Canary Islands
  - Research Site, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Research Site, Santander, Cantabria
  - Hospital Nuestra Señora de Sonsoles, Ávila, Castille and León
  - Hospital Universitario Río hortega de Valladolid, Valladolid, Castille and León
  - Research Site, Valladolid, Castille and León
  - Hospital Germans Tries i Pujol, Badalona, Catalonia
  - Research Site, Badalona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Research Site, Barcelona, Catalonia
  - Hospital Sant Pau, Barcelona, Catalonia
  - Hospital Valle Hebrón, Barcelona, Catalonia
  - Hospital de Bellvitge, Barcelona, Catalonia
  - Hospital Mutua de Terrassa, Terrassa, Catalonia
  - Hospital Infanta Cristina Badajoz, Badajoz, Extremadura
  - Hospital Universitario de Ourense, Ourense, Galicia
  - Hospital Universitario de Pontevedra, Pontevedra, Galicia
  - Research Site, Móstoles, Madrid
  - Hospital Santa Lucía, Cartagena, Murcia, Murcia
  - Hospital General de Alicante, Alicante, Valencia
  - Hospital Clínico Valencia, Valencia, Valencia
  - Hospital General Valencia, Valencia, Valencia
  - Hospital La Fe Valencia, Valencia, Valencia
  - Research Site, Alicante
  - Research Site, Ávila
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Cuesta
  - Research Site, Huelva
  - Research Site, Jaén
  - Hospital La Princesa, Madrid
  - Research Site, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital de 12 Octubre, Madrid
  - Hospital Universitario Puerta del Hierro, Madrid
  - Hospital de Móstoles, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Murica
  - Research Site, Ourense
  - Research Site, Pontevedra
  - Research Site, Terrassa
  - Research Site, Valencia
  - Research Site, Zaragoza
  - Hospital Clínico de Zaragoza, Zaragoza, Áragon
  - Hospital Miguel Servet, Zaragoza, Áragon

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Expanded Access for CC-10004 — https://clinicaltrials.gov/ct2/show/NCT03539419?term=CC-10004-PSOR-017&rank=1